CLINICAL TRIAL: NCT02449720
Title: The Effect of Intraperitoneal Local Anaesthetic on Functional Recovery Following Bowel Resection: A Prospective Randomised Blinded Trial
Brief Title: Intraperitoneal Local Anaesthetic in Bowel Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Royal Adelaide Hospital (Other)
Collaborators: University of Adelaide (Other); University of South Australia (Other); Saint Andrew's Hospital (Unknown); Calvary North Adelaide Hospital (Unknown)
Responsible Party: Principal Investigator, Dr Jaime A Duffield, Colorectal Surgical Unit Research Registrar, Royal Adelaide Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 150219
Record Dates: First submitted 2015-04-28; First posted 2015-05-20 (Estimated); Last update posted 2017-03-27 (Actual); Status verified 2017-03

CONDITIONS: Colorectal Disorders
Keywords: intraperitoneal; ropivacaine; bowel resection; local anaesthetic; recovery
MeSH Terms: interventions — Ropivacaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Laparoscopic Bowel Surgery: IPLA (Active Comparator): Participants will undergo laparoscopic bowel surgery. Both on entry into the abdominal cavity and prior to dissection and post-operation but prior to closure of abdominal wall a 50 ml loading dose of IPLA (0.2% Ropivacaine) solution will be distributed throughout the abdomen. Following these bolus doses an ON-Q Painbuster continuous infusion pump will be placed in close proximity to the operative region of greatest dissection and a 10ml/hr intraperitoneal infusion of IPLA (0.2% Ropivacaine, 20mg/hr) solution commenced immediately post-operation and continued for 48 hrs without disruption.
  Interventions: Drug: Ropivacaine
- Laparoscopic Bowel Surgery: Control (Placebo Comparator): Participants will undergo laparoscopic bowel surgery. Both on entry into the abdominal cavity and prior to dissection and post-operation but prior to closure of abdominal wall a 50 ml loading dose of Control (0.9% Saline, 20mg/hr) solution will be distributed throughout the abdomen. Following these bolus doses an ON-Q Painbuster continuous infusion pump will be placed in close proximity to the operative region of greatest dissection and a 10ml/hr intraperitoneal infusion of Control (0.9% Saline, 20mg/hr) solution commenced immediately post-operation and continued for 48 hrs without disruption.
  Interventions: Drug: 0.9% Saline
- Open Bowel Surgery: IPLA (Active Comparator): Participants will undergo open bowel surgery. Both on entry into the abdominal cavity and prior to dissection and post-operation but prior to closure of abdominal wall a 50 ml loading dose of IPLA (0.2% Ropivacaine) solution will be distributed throughout the abdomen. Following these bolus doses an ON-Q Painbuster continuous infusion pump will be placed in close proximity to the operative region of greatest dissection and a 10ml/hr intraperitoneal infusion of IPLA (0.2% Ropivacaine, 20mg/hr) solution commenced immediately post-operation and continued for 48 hrs without disruption.
  Interventions: Drug: Ropivacaine
- Open Bowel Surgery: Control (Placebo Comparator): Participants will undergo open bowel surgery. Both on entry into the abdominal cavity and prior to dissection and post-operation but prior to closure of abdominal wall a 50 ml loading dose of Control (0.9% Saline, 20mg/hr) solution will be distributed throughout the abdomen. Following these bolus doses an ON-Q Painbuster continuous infusion pump will be placed in close proximity to the operative region of greatest dissection and a 10ml/hr intraperitoneal infusion of Control (0.9% Saline, 20mg/hr) solution commenced immediately post-operation and continued for 48 hrs without disruption.
  Interventions: Drug: 0.9% Saline

INTERVENTIONS:
Drug: Ropivacaine — Intraperitoneal instillation and infusion
  Other Names: Naropin
  Arms: Laparoscopic Bowel Surgery: IPLA; Open Bowel Surgery: IPLA
Drug: 0.9% Saline — Intraperitoneal instillation and infusion
  Other Names: Normal Saline
  Arms: Laparoscopic Bowel Surgery: Control; Open Bowel Surgery: Control

SUMMARY:
This study will evaluate the addition of a local anaesthetic infusion into the abdomen to patient controlled analgesia in the management of postoperative pain and recovery after bowel surgery. Half of the patients will have an infusion of a local anaesthetic called ropivacaine and half will have an infusion of placebo in addition to their normal pain relief.

DETAILED DESCRIPTION:
The purpose of this randomised controlled blinded trial is to determine the effectiveness in every day practice of intraperitoneal local anaesthetic (IPLA) infusion on postoperative recovery following bowel resection in an optimised Enhanced Recovery After Surgery (ERAS) setting.

The investigators hypothesise that, in an optimised ERAS setting, intraperitoneal instillation and infusion of the local anaesthetic ropivacaine to the site of maximal visceral dissection for 48 hrs will result in an improved functional postoperative recovery following both open and laparoscopic bowel surgery.

This research will provide evidence to allow recommendation on the routine inclusion of IPLA into the multimodal analgesia component of ERAS programs for bowel surgery.

ELIGIBILITY:
Inclusion Criteria:

* The study population will include adults from the Central Adelaide Local Health network catchment area, South Australia.
* Patients known to the Colorectal Surgical Unit who have provided informed consent to undergo elective large bowel resection for any indication or undergoing reversal of Hartmann's Procedure will be invited to participate in this study.
* Potential participants will then be provided with an Information Sheet and encouraged to take the time to read it, discuss it with anyone they like, and ask any questions they have prior to deciding if they wish to participate. They will be reassured that participation is voluntary and there is no disadvantage to them if they decide not to participate.
* After obtaining informed consent, eligibility for inclusion will be determined based on health questions and blood results.

Exclusion Criteria:

* Under 18 years of age or over age 90.
* Allergy to local anaesthetic.
* Underlying medical conditions requiring deviation from the proposed anaesthetic protocol i.e., use of spinal or epidural anaesthesia rather than general anaesthesia.
* American Society of Anesthesiologists (ASA) >=4 due to the higher likelihood or morbidity and mortality, which may confound resulting data.
* Severe underlying cardiovascular disease including conduction abnormalities, ischaemic heart disease or congestive heart failure, or use of amiodarone as a regular medication due to a higher risk or cardiac arrest under general anaesthetic or during use of local anaesthesia.
* Chronic Renal Failure (CRF) Stage 3 (GFR > 60 based on two samples a minimum 90d apart).
* The pharmacokinetics of ropivacaine is not affected by renal failure although the renal clearance of its main metabolite (S)-2',6'-pipecoloxylidide (PPX) correlates with creatinine clearance, non-renal clearance compensates for reduced renal clearance in most patients.
* GFR will be calculated using the Cockcroft Gault equation for creatinine clearance (CrCl) : CrCl ml/min = [140-age(years)] x bodyweight (kg) / R x serum creatinine (micromol/L)
* R = 0.815 for males, 0.85 for females
* Hepatic dysfunction of Child-Pugh class B or C. Patients with end-stage liver disease have about a 60% lower mean ropivacaine clearance than healthy subjects and are thus expected to have over two-fold higher steady-state ropivacaine plasma concentrations during a continuous ropivacaine infusion.
* Concurrent or recent (within 3 months) use of fluvoxamine, enoxacin, ketoconazole, or cimetidine. These are potent CYP (cytochrome P450) 1A2, 2E1, or 3A4 inhibitors that have been shown to reduce ropivacaine clearance in vivo or in in vitro models. Potential participants concurrently using other potent CYP1A2, 2E1, or 3A4 inhibitors, where it is unclear if there is an effect on ropivacaine clearance, will be included or excluded from the study at the discretion of their study specialist anaesthetist.
* Abdominal-perineal resections (APR) due to the greater area of dissection and skin incision which will increase the level of baseline somatic pain felt by a patient.
* Requirement for postoperative drain in-situ, as this will drain the experimental solution out of the abdomen.
* Preoperative systemic steroid dependence due to derangement of the inflammatory response.
* Preoperative chronic pain illness including fibromyalgia, chronic regional pain syndrome, chronic fatigue syndrome, non specific chronic pain requiring daily opiate use, and history of alcohol or drug dependence due to the impact these have on subjective interpretation of pain and tolerance to opioid requiring significantly higher dosing regimens.
* Inability to consent or complete data scores in the study questionnaires due to cognitive impairment and/or language barrier.
* Pregnancy or breastfeeding.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2015-05; Primary Completion 2016-06 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change from Baseline of the Surgical Recovery Scale to Day 45 | Baseline (preoperative), and postoperative days 1, 3, 7, 30 and 45
  The postoperative domains of recovery of fatigue, and the post-discharge return to normal functioning in both cognition (concentration) and activities of daily living will be assessed using the Surgical Recovery Scale, previously validated for use following bowel surgery.

SECONDARY OUTCOMES:
Change in Pain Over Time to Day 7 (Subjective) | At postoperative hours 3, 6, 12, 24, 48, and 72, and at day 7
  Postoperative pain at rest and with movement (defined as coughing) will be evaluated using a 100mm Visual Analogue Scale with the end-points labelled "no pain" and "the worst possible pain" for each of: I. somatic pain (incisional pain in the abdominal wall that the patient can touch) II. visceral pain (deep, dull, inside the abdomen) III. shoulder tip pain
Change in Pain Over Time to day 3 (Objective) | Postoperative day 1, 2, and 3
  Total opioid analgesia use during the postoperative day 1, 2, and 3 prior to discharge will be recorded and quantified using the Mean Equivalent Daily Dose (MEDD) method. Initially this will be parenteral fentanyl consumption, recorded daily in the patient controlled analgesia (PCA) device until removal of PCA. Then this will be prn tramadol, or other opioid as charted, until discharge.
  Time to first PCA button press, and the number of PCA button presses will also be recorded as sometimes patients would like more analgesia than the PCA is able to administer.
Recovery of Normal Bowel Function | Inpatient postoperative period (variable), and expected duration of 3-7 days.
  Time to tolerating oral diet and to first postoperative flatus, and bowel motion will be recorded. Post-operative antiemetic use will be recorded, as will number of episodes of vomiting. The length of time requiring postoperative intravenous fluid will be recorded. The requirement for insertion of naso-gastric tube will be recorded.
Time to Readiness for Discharge | up to 30 days
  The time to readiness for discharge (TRD) is a validated measurement of short-term recovery after colorectal surgery. TRD and actual length of stay (LOS) will be recorded.
  Discharge criteria will be defined as
  1. Passage of flatus or bowel motion, tolerance of oral diet and absence of nausea and vomiting.
  2. Mobilisation back to baseline function.
  3. Analgesia requirement managed with oral tablets only.
  4. Willingness to be discharged home. Readmission, defined as unplanned return to hospital within 30 day and requiring an overnight admission, will be recorded.
  Total hospital stay will be recorded as LOS + readmission LOS.
Operative Complications | 30 days post operation
  All complications that occur within a 30d postoperative period will be recorded. Complications will be recorded and graded using the Clavien-Dindo classification system.

CONTACTS AND LOCATIONS:
Overall Officials: Jaime A Duffield, BMBS PhD, Principal Investigator — Royal Adelaide Hospital, Colorectal Surgical Unit Research Registrar
Locations (1):
- Royal Adelaide Hospital, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Paddison JS, Sammour T, Kahokehr A, Zargar-Shoshtari K, Hill AG. Development and validation of the Surgical Recovery Scale (SRS). J Surg Res. 2011 May 15;167(2):e85-91. doi: 10.1016/j.jss.2010.12.043. Epub 2011 Jan 31. PMID 21392804
- [Result] Kahokehr A, Sammour T, Zargar Shoshtari K, Taylor M, Hill AG. Intraperitoneal local anesthetic improves recovery after colon resection: a double-blinded randomized controlled trial. Ann Surg. 2011 Jul;254(1):28-38. doi: 10.1097/SLA.0b013e318221f0cf. PMID 21670611
- [Derived] Duffield JA, Thomas ML, Moore JW, Hunter RA, Wood C, Gentili S, Lewis M. Intraperitoneal Local Anesthetic Instillation and Postoperative Infusion Improves Functional Recovery Following Colectomy: A Randomized Controlled Trial. Dis Colon Rectum. 2018 Oct;61(10):1205-1216. doi: 10.1097/DCR.0000000000001177. PMID 30192329